CLINICAL TRIAL: NCT05627895
Title: A Feasibility Study of fMRI-neurofeedback in Parkinson's Disease
Brief Title: Brain Self-regulation for Parkinson's
Acronym: Brain-REG
Status: Completed | Type: Observational
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: NL82024.068.22
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Basal-ganglia fMRI Neurofeedback
Keywords: Neurofeedback; Self-regulation; Functional MRI
MeSH Terms: conditions — Self-Control | interventions — Neurofeedback

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient cohort: All patients will undergo both the SMA and the basal ganglia condition
  Interventions: Other: Neurofeedback

INTERVENTIONS:
Other: Neurofeedback — Participants will be shown their brain activity measured in real-time using an MRI scanner. They can then use mental strategies, such as imagination to influence and regulate this activity.
  Other Names: fMRI based neurofeedback; Self-regulation of brain activity using neurofeedback

SUMMARY:
To investigate feasibility of basal-ganglia regions as fMRI-neurofeedback targets in Parkinson's patients and evaluate self-regulation success

DETAILED DESCRIPTION:
This is a single-group proof of mechanism study of Parkinson's Disease (PD) patients receiving neurofeedback (NF) training using supplementary motor area (SMA) and basal ganglia as target areas. At the start of the screening session, consent will be taken. Subsequently, the screening assessment will be performed to determine inclusion and exclusion criteria. After inclusion in the study has been established, the NF sessions at the MRI scanner will be scheduled. The participants will be invited for up to three NF sessions. This will total up to a maximum of four visits, one for screening and up to three for the NF sessions. Due to the feasibility nature of the study, the optimal number of sessions for the patient cohort to learn the NF regulation is unknown. Therefore, flexibility has been introduced in the design to facilitate learning in case it is necessary. The NF training is modelled on the investigators' previous work.

Each NF session will consist of one anatomical scan, one localizer run, and four functional NF runs. The localizer run will be used to identify individualized brain activation patterns in the participants. Each NF run is a measurement sequence that will consist of ten blocks: five regulation blocks and five rest blocks. The participants will be asked to upregulate (increase) their brain activity, which will be displayed on a thermometer bar, during the regulation blocks. During the rest blocks, the participants will be asked to relax. The study will employ a crossover design with two conditions. In one condition the participants will receive feedback on the thermometer bar from the SMA region and in the second condition the participants will receive feedback from the basal ganglia region. Two of the NF runs will be with the SMA condition and two will be with the basal ganglia condition. Both runs in each condition will take place consecutively, i.e., either the first two runs will be SMA and the second two runs will be basal ganglia or vice versa. The sessions will be counter balanced.

At the last NF session, a post-training assessment will be conducted during which the participants will be debriefed about the study. NF is an individualized training method, and therefore, individual differences in learning success are expected during the study, which can lead to different expectations from the subjects. However, since this is an investigation of the feasibility of the approach, all forms of performance are useful datapoints and participants will be debriefed about their valuable contribution to make sure that no outcome is conceived as negative.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease (see 4.1) according to Movement Disorder Society (MDS) clinical diagnostic criteria (Postuma et al., 2015).
* Disease stage 1-3 according to the Hoehn and Yahr Scale

Exclusion Criteria:

* Exclusion criteria for MRI (e.g., cardiac pacemaker, certain metallic implants)
* History of psychotic disorder, bipolar disorder, or psychotic depression
* Current use of illegal drugs (any in the last four weeks)
* Current excessive alcohol consumption that interferes with daily functioning
* Advanced cognitive impairment (MoCA <24) or dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease as per inclusion/ exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of basal-ganglia neurofeedback training (fMRI analysis) | Measurements will be recorded at each MRI session (approx. 1 week intervals after screening and inclusion)
  We will be investigating the ability of the basal ganglia to be used as a neurodeedback target for self-regulation in PD patients. To determine the ability of the basal ganglia to be recruited in the neurofeedback training, we will look at the T-contrast of all basal ganglia regulation blocks vs all baseline blocks in all the runs where basal ganglia was the target region.

SECONDARY OUTCOMES:
Performance of basal-ganglia neurofeedback training (fMRI analysis) | Measurements will be recorded at each MRI session (approx. 1 week intervals after screening and inclusion)
  To determine the performance of basal ganglia self-regulation, we will employ a T-contrast of all runs with the basal ganglia as the target region versus all the runs with the SMA as the target region. Additionally, we will assess whole-brain activation changes in the basal ganglia runs to determine specificity of the neurofeedback training. This can give us insight into which brain networks contribute mechanistically to the training and if any of the training performance can be attributed to other factors, such as physiological measures, as compared to neurofeedback self-regulation.

CONTACTS AND LOCATIONS:
Overall Officials: David EJ Linden, Prof., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Emmert K, Kopel R, Sulzer J, Bruhl AB, Berman BD, Linden DEJ, Horovitz SG, Breimhorst M, Caria A, Frank S, Johnston S, Long Z, Paret C, Robineau F, Veit R, Bartsch A, Beckmann CF, Van De Ville D, Haller S. Meta-analysis of real-time fMRI neurofeedback studies using individual participant data: How is brain regulation mediated? Neuroimage. 2016 Jan 1;124(Pt A):806-812. doi: 10.1016/j.neuroimage.2015.09.042. Epub 2015 Sep 28. PMID 26419389
- [Background] Hamilton JP, Glover GH, Bagarinao E, Chang C, Mackey S, Sacchet MD, Gotlib IH. Effects of salience-network-node neurofeedback training on affective biases in major depressive disorder. Psychiatry Res Neuroimaging. 2016 Mar 30;249:91-6. doi: 10.1016/j.pscychresns.2016.01.016. Epub 2016 Jan 19. PMID 26862057
- [Background] Jaeckle T, Williams SCR, Barker GJ, Basilio R, Carr E, Goldsmith K, Colasanti A, Giampietro V, Cleare A, Young AH, Moll J, Zahn R. Self-blame in major depression: a randomised pilot trial comparing fMRI neurofeedback with self-guided psychological strategies. Psychol Med. 2023 May;53(7):2831-2841. doi: 10.1017/S0033291721004797. Epub 2021 Dec 2. PMID 34852855
- [Background] Johnston SJ, Boehm SG, Healy D, Goebel R, Linden DE. Neurofeedback: A promising tool for the self-regulation of emotion networks. Neuroimage. 2010 Jan 1;49(1):1066-72. doi: 10.1016/j.neuroimage.2009.07.056. Epub 2009 Jul 29. PMID 19646532
- [Background] Linden DE. Neurofeedback and networks of depression. Dialogues Clin Neurosci. 2014 Mar;16(1):103-12. doi: 10.31887/DCNS.2014.16.1/dlinden. PMID 24733975
- [Background] Linden DE, Habes I, Johnston SJ, Linden S, Tatineni R, Subramanian L, Sorger B, Healy D, Goebel R. Real-time self-regulation of emotion networks in patients with depression. PLoS One. 2012;7(6):e38115. doi: 10.1371/journal.pone.0038115. Epub 2012 Jun 4. PMID 22675513
- [Background] MacDuffie KE, MacInnes J, Dickerson KC, Eddington KM, Strauman TJ, Adcock RA. Single session real-time fMRI neurofeedback has a lasting impact on cognitive behavioral therapy strategies. Neuroimage Clin. 2018 Jun 9;19:868-875. doi: 10.1016/j.nicl.2018.06.009. eCollection 2018. PMID 29922575
- [Background] Mehler DMA, Sokunbi MO, Habes I, Barawi K, Subramanian L, Range M, Evans J, Hood K, Luhrs M, Keedwell P, Goebel R, Linden DEJ. Targeting the affective brain-a randomized controlled trial of real-time fMRI neurofeedback in patients with depression. Neuropsychopharmacology. 2018 Dec;43(13):2578-2585. doi: 10.1038/s41386-018-0126-5. Epub 2018 Jun 23. PMID 29967368
- [Background] Mehler DMA, Williams AN, Krause F, Luhrs M, Wise RG, Turner DL, Linden DEJ, Whittaker JR. The BOLD response in primary motor cortex and supplementary motor area during kinesthetic motor imagery based graded fMRI neurofeedback. Neuroimage. 2019 Jan 1;184:36-44. doi: 10.1016/j.neuroimage.2018.09.007. Epub 2018 Sep 8. PMID 30205210
- [Background] Paret C, Zaehringer J, Ruf M, Ende G, Schmahl C. The orbitofrontal cortex processes neurofeedback failure signals. Behav Brain Res. 2019 Sep 2;369:111938. doi: 10.1016/j.bbr.2019.111938. Epub 2019 May 6. PMID 31071348
- [Background] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316
- [Background] Sitaram R, Ros T, Stoeckel L, Haller S, Scharnowski F, Lewis-Peacock J, Weiskopf N, Blefari ML, Rana M, Oblak E, Birbaumer N, Sulzer J. Closed-loop brain training: the science of neurofeedback. Nat Rev Neurosci. 2017 Feb;18(2):86-100. doi: 10.1038/nrn.2016.164. Epub 2016 Dec 22. PMID 28003656
- [Background] Skottnik L, Linden DEJ. Mental Imagery and Brain Regulation-New Links Between Psychotherapy and Neuroscience. Front Psychiatry. 2019 Oct 30;10:779. doi: 10.3389/fpsyt.2019.00779. eCollection 2019. PMID 31736799
- [Background] Skottnik L, Sorger B, Kamp T, Linden D, Goebel R. Success and failure of controlling the real-time functional magnetic resonance imaging neurofeedback signal are reflected in the striatum. Brain Behav. 2019 Mar;9(3):e01240. doi: 10.1002/brb3.1240. Epub 2019 Feb 20. PMID 30790474
- [Background] Subramanian L, Hindle JV, Johnston S, Roberts MV, Husain M, Goebel R, Linden D. Real-time functional magnetic resonance imaging neurofeedback for treatment of Parkinson's disease. J Neurosci. 2011 Nov 9;31(45):16309-17. doi: 10.1523/JNEUROSCI.3498-11.2011. PMID 22072682
- [Background] Subramanian L, Morris MB, Brosnan M, Turner DL, Morris HR, Linden DE. Functional Magnetic Resonance Imaging Neurofeedback-guided Motor Imagery Training and Motor Training for Parkinson's Disease: Randomized Trial. Front Behav Neurosci. 2016 Jun 8;10:111. doi: 10.3389/fnbeh.2016.00111. eCollection 2016. PMID 27375451
- [Background] Young KD, Siegle GJ, Zotev V, Phillips R, Misaki M, Yuan H, Drevets WC, Bodurka J. Randomized Clinical Trial of Real-Time fMRI Amygdala Neurofeedback for Major Depressive Disorder: Effects on Symptoms and Autobiographical Memory Recall. Am J Psychiatry. 2017 Aug 1;174(8):748-755. doi: 10.1176/appi.ajp.2017.16060637. Epub 2017 Apr 14. PMID 28407727
- [Background] Zahn R, Weingartner JH, Basilio R, Bado P, Mattos P, Sato JR, de Oliveira-Souza R, Fontenelle LF, Young AH, Moll J. Blame-rebalance fMRI neurofeedback in major depressive disorder: A randomised proof-of-concept trial. Neuroimage Clin. 2019;24:101992. doi: 10.1016/j.nicl.2019.101992. Epub 2019 Aug 25. PMID 31505367